CLINICAL TRIAL: NCT06273982
Title: Behavioral Telehealth in Low-resource Primary Care Settings for Anxiety and Depression in Youth: A Randomized Effectiveness-implementation Study
Brief Title: Behavioral Telehealth in Low-resource Primary Care Settings for Anxiety and Depression in Youth
Acronym: STEP-UP
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Collaborators: Kaiser Permanente (Other); OCHIN, Inc. (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HS-2023-0281-SMT; 1R01MH131698 (NIH)
Record Dates: First submitted 2024-02-15; First posted 2024-02-23 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Depression, Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STEP-UP (Experimental)
  Interventions: Behavioral: STEP-UP (transdiagnostic behavioral therapy for pediatric anxiety and depression)
- ARC (Active Comparator)
  Interventions: Behavioral: ARC (assisted referral to community care)

INTERVENTIONS:
Behavioral: STEP-UP (transdiagnostic behavioral therapy for pediatric anxiety and depression) — STEP-UP consists of 8 to 12 sessions of behavioral therapy for anxiety and / or depression. Skills taught include relaxation, problem solving, and exposure / behavioral activation.
  Other Names: Brief Behavioral Therapy (BBT) for pediatric anxiety and depression
  Arms: STEP-UP
Behavioral: ARC (assisted referral to community care) — ARC consists of referral to community mental health treatment-as-usual. Families are provided psychoeducation about anxiety and depression and the benefits of treatment, lists of local community providers, and a problem-solving discussion about obstacles to obtaining care.
  Arms: ARC

SUMMARY:
The goal of this clinical trial is to test a brief, behavioral telehealth treatment program (STEP-UP) for depression and anxiety in youths (age 8-16 years old). Youths and families will be recruited through participating community health centers and will be randomly assigned to either: (a) receive STEP-UP care from providers at their health center or (b) be referred to care from local community mental health clinicians. Youth and families will be interviewed before treatment starts, 16 weeks later, and 24 weeks later to assess how youth are feeling. The main question the study aims to answer is whether STEP-UP improves youths functioning in daily life, anxiety symptoms, and depression symptoms. Researchers will compare STEP-UP to referral to community treatment-as-usual mental health services to see if STEP-UP is more effective.

ELIGIBILITY:
Inclusion Criteria:

* Youth is a patient in a participating community health center.
* Youths meet criteria for clinically significant anxiety and / or depression as indexed at baseline assessment by either:

  * research diagnosis of anxiety (Social Anxiety Disorder, Generalized Anxiety Disorder, Separation Anxiety Disorder) and / or depressive disorder (Major Depressive Disorder, Persistent Depressive Disorder).
  * scores in the clinically elevated range on a standardized anxiety and / or depression symptom measure .
* Youth lives with a legal guardian (hereafter referred to as "parent") >= 50% of the time who consents to study participation.
* Youth speaks English.
* Parent speaks English or Spanish.

Exclusion Criteria:

* Youth requires alternate treatment as indexed by:

  * current clinically significant Post-Traumatic Stress Disorder symptoms (meets diagnostic criteria in research interview and / or scores in the clinically elevated range on a standardized symptom measure) at baseline.
  * current suicidal ideation with plan at baseline and / or suicidal behavior within the last year.
  * current substance dependence at baseline.
  * experience of physical or sexual abuse within the six months prior to baseline.
  * parent /guardian does not identify anxiety and / or depression as a treatment priority at baseline.
* Youth is in an active, alternate psychosocial intervention for anxiety or depression that would be concurrent with study participation.
* Youth is on an unstable regimen of psychotropic medication (i.e., receives medication but has not been at a stable dose for at least 8 weeks, or if medication has been discontinued for less than 4 weeks) at baseline.
* Youth is receiving lithium or and anti-psychotic medication at baseline.
* Youth is placed in a special education program for greater than 50% of the school day and / or youth school placement is below the second-grade level at baseline.
* Youth is placed in foster care at baseline.

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 220 (Estimated)
Dates: Start 2024-07-09 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Children's Global Assessment Scale (CGAS) | Measured at baseline (Week 0) and follow-up assessments (Week 16 and Week 32)
  Interviewer-rated youth functioning. Scores range from 1 to 100, and higher score indcate superior functioning.
Pediatric Anxiety Rating Scale (PARS) | Measured at baseline (Week 0) and follow-up assessments (Week 16 and Week 32). The PARS total severity score ranges from 0 to 30, with higher scores indicating greater anxiety severity.
  Interviewer-rated symptoms of anxiety disorders, combining parent and youth report
Children's Depression Rating Scale -- Revised (CDRS-R) | Measured at baseline (Week 0) and follow-up assessments (Week 16 and Week 32). The CDRS-R total severity score ranges from 17 to 113, with higher scores indicating greater depression symptom severity.
  Interviewer rated symptoms of depressive disorders, combining parent and youth report

CONTACTS AND LOCATIONS:
Overall Officials: V. Robin Weersing, PhD, Principal Investigator — San Diego State University; Frances Lynch, PhD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Center for Health Research, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes